CLINICAL TRIAL: NCT02438813
Title: CONTOUR: Condition of Submental Fullness and Treatment Outcomes Registry (A Registry of Submental Fullness, Treatment Options Administered, and Associated Outcomes)
Brief Title: Condition of Submental Fullness and Treatment Outcomes Registry
Acronym: CONTOUR
Status: Completed | Type: Observational
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CONTOUR
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Submental Fullness
MeSH Terms: interventions — Deoxycholic Acid; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: All enrolled participants who signed informed consent whether or not they elected to receive treatment as per standard of care in clinical practice for submental fat (SMF). Treatments for SMF included: ATX1-101, Surgical Procedures, Laser Liposuction, Energy Devices or Other Treatments.
  Interventions: Drug: Deoxycholic acid; Procedure: Surgical Procedures; Procedure: Laser Liposuction; Device: Energy Devices; Other: Other Treatments

INTERVENTIONS:
Drug: Deoxycholic acid — Deoxycholic acid (ATX-101) injection as the treatment of SMF as per standard of care in clinical practice.
  Other Names: ATX-101; KYBELLA
Procedure: Surgical Procedures — Surgical procedures for treatment of SMF as per standard of care in clinical practice.
Procedure: Laser Liposuction — Laser Liposuction for the treatment of SMF as per standard of care in clinical practice..
Device: Energy Devices — Energy Devices for the treatment of SMF as per standard of care in clinical practice.
Other: Other Treatments — Other treatments for SMF as per standard of care in clinical practice.

SUMMARY:
The primary objective of this registry is to develop a comprehensive understanding of the condition of submental (SM) fullness due to submental fat (SMF), how it is treated in current clinical practice, and the risks and benefits associated with its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, aged 18 years and above, presenting with SM fullness due to the accumulation of unwanted SMF, and considered by their treating physician to be a candidate to receive treatment of SM fullness by reduction of SMF, if the patient decides
* Signed informed consent by the patient, obtained before any study-related activities are undertaken
* Willing to complete all patient assessment questionnaires
* Signed release form by the patient, permitting abstraction of the patient's medical records at baseline and during participation in the registry

Exclusion Criteria:

* Severe skin laxity, defined as superficial wrinkling, loose skin separated from deeper neck structures, and/or marked skin redundancy (draping and/or sagging), per the physician's judgment
* Any other cause of fullness in the SM area (eg, thyroid enlargement, cervical adenopathy) other than localized SMF
* Participating in an interventional clinical study, currently or within 30 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients considering treatment to reduce SMF will be recruited from practices that see a large number of aesthetic patients with a variety of issues, including SMF.
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rina Patel, MS, CCRA, Study Director — Allergan
Locations (95):
- United States (84):
  - Skin Spectrum LLC, Tucson, Arizona
  - John Joseph, MD, Beverly Hills, California
  - The Roxbury Institute, Beverly Hills, California
  - Brian M Kinney, MD Inc, Beverly Hills, California
  - Bella Skin Institute, Calabasas, California
  - Jerome R Potozkin MD, Danville, California
  - Kathleen L Behr, Fresno, California
  - Ocdermatology Lorrie Klein, Laguna Niguel, California
  - Westside Aesthetics, Los Angeles, California
  - Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California
  - Batniji Facial Plastic Surgery, Newport Beach, California
  - Steve Yoelin, M.D. Medical Associates, Inc., Newport Beach, California
  - Teleos Plastic Surgery &. Radiance Medical Group Inc, Pasadena, California
  - Laser And Skin Surgery Center Of Northern California, Sacramento, California
  - Dermatology Cosmetic Laser Medical Associates of La JollaInc, San Diego, California
  - FacesPlus, San Diego, California
  - Goldman Butterwick Fitzpatrick Groff And Fabi Cosmetic Laser, San Diego, California
  - The Maas Clinic - San Francisco, San Francisco, California
  - Bay Area Cosmetic Dermatology Kathleen M Welsh Md, San Francisco, California
  - Vic A Narurkar MD APC, San Francisco, California
  - Grossman Dermatology, Santa Monica, California
  - Art Of Skin MD, Solana Beach, California
  - Moradi Md, Vista, California
  - Practice Dr Mary Lynn Moran, Woodside, California
  - AboutSkin Dermatology and Dermsurg, Greenwood Village, Colorado
  - Wa Institute Dermatologic Laser Surg, Washington D.C., District of Columbia
  - Sanctuary Medical Aesthetic Center, Boca Raton, Florida
  - Steven Fagien, MD, PA, Boca Raton, Florida
  - Skin Care Research, Inc, Boca Raton, Florida
  - Susan H Weinkle Md, Bradenton, Florida
  - Skin Research Institute, Coral Gables, Florida
  - The Miami Institute, Miami, Florida
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Center For Sight, Sarasota, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Carmen Kavali, Atlanta, Georgia
  - John Connors Plastic Surgery, Atlanta, Georgia
  - DeNova Research, Chicago, Illinois
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Coleman Center For Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - Lupo Center for Aesthetic and General Dermatology, New Orleans, Louisiana
  - Facial Plastic Surgical Center, Baltimore, Maryland
  - Dermatologic Surgery Center of Washington LLC, Chevy Chase, Maryland
  - Callender Center for Clinical Research, LLC, Glenn Dale, Maryland
  - Maryland Laser Skin & Vein Inst, Hunt Valley, Maryland
  - Lawrence Green MD LLC, Rockville, Maryland
  - Ranella Hirsch, Cambridge, Massachusetts
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Dermatology Partners, Wellesley, Massachusetts
  - Boyd, Birmingham, Michigan
  - United Skin Specialists LTD, Edina, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Skin Specialists, P.C., Omaha, Nebraska
  - Practice Dr Angela Beckford, Hackensack, New Jersey
  - Image Dermatology P.C., Montclair, New Jersey
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Forest Hills Dermatology Group, Forest Hills, New York
  - The Center For Dermatology Cosmetic And Laser Surgery, Mount Kisco, New York
  - Beth Israel Medical Center, New York, New York
  - Doris Day Pc, New York, New York
  - New York Cosmetic, Skin and Laser Surgery Center (NYC), New York, New York
  - JUVA Skin and Laser Center, New York, New York
  - Marmur Medical, New York, New York
  - New York Laser and Skin Care, New York, New York
  - Luxurgery NYC, New York, New York
  - Sadick Research Group, New York, New York
  - Marina I Peredo M.D., P.C., Smithtown, New York
  - Mariwalla Dermatology, West Islip, New York
  - Finn Facial Plastics, Chapel Hill, North Carolina
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Oregon Health And Science University Hospital, Portland, Oregon
  - Main Line Center for Laser Surgery, Ardmore, Pennsylvania
  - Plaza Surgical Center, Bala-Cynwyd, Pennsylvania
  - Dermatologic SurgiCenter, Drexel Hill, Pennsylvania
  - Brian S. Biesman, M.D., Nashville, Tennessee
  - Westlake Dermatology And Cosmetic Surgery, Austin, Texas
  - Bellaire Dermatology Associates (BDA), Bellaire, Texas
  - Research Across America, Plano, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Gateway Aesthetic Institute & Laser Center, Salt Lake City, Utah
  - Hema A Sundaram MDPA, Fairfax, Virginia
  - Naficy Plastic Surgery And Rejuvenation Center, Bellevue, Washington
  - Premier Clinical Research, Spokane, Washington
- Canada (11):
  - Dr. Shannon Humphrey, Inc., Vancouver, British Columbia
  - Pacific Dermaesthetics, Vancouver, British Columbia
  - Project Skin Vancouver, Vancouver, British Columbia
  - Dr. Jean Carruthers Cosmetic Surgey Inc., Vancouver, B. C., British Columbia
  - North York General Hospital, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Compass Dermatology, Toronto, Ontario
  - Sweat Clinics of Canada, Toronto, Ontario
  - Bertucci MedSpa, Inc., Woodbridge, Ontario
  - Medime Institut de medecine esthetique, Montreal, Quebec
  - Dr. Nikolis, Mount Royal, Quebec

REFERENCES:
- [Derived] Palm MD, Schlessinger J, Callender VD, Fagien S, Beer K, Magante S, Sangha S. Final Data from the Condition of Submental Fullness and Treatment Outcomes Registry (CONTOUR). J Drugs Dermatol. 2019 Jan 1;18(1):40-48. PMID 30681793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 1029
Received Treatment for SMF | 676
Did Not ReceiveTreatment for SMF | 353
Completed | 504
Not Completed | 525
Not completed — Patient Decision | 59
Not completed — Patient Lost to Follow-Up | 137
Not completed — Study Ended by Sponsor | 80
Not completed — Patients Not Treated/No EOT Visit | 249

BASELINE CHARACTERISTICS:
Population: Enrolled Participants include all participants who signed informed consent whether or not they elected to receive treatment.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1029
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.30)
Age, Customized [Number; unit: participants]
  18 to 30 years | 81
  31 to 50 years | 427
  51 to 65 years | 413
  >65 years | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 883
  Male | 146

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event is any undesirable medical occurrence or worsening of an existing condition that occurs after SMF reduction treatment, irrespective of whether the event is considered treatment related. A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving treatment.
Time Frame: Up to 19 Months
Population: Safety Population included all participants who received at least one treatment. Participants may have received more than one treatment.
Measure: Number; unit: percentage of participants
Groups:
- Deoxycholic Acid (ATX-101): Deoxycholic acid injection (ATX-101) as treatment for SMF as per standard of care.
- Surgical: Surgical procedures for the treatment of SMF as per standard of care in clinical practice.
- Laser Liposuction: Laser Liposuction for treatment of SMF as per standard of care in clinical practice.
- Energy Devices: Energy Devices as treatment for SMF as per standard of care in clinical practice.
- Other Treatments: Other Treatments for treatment of SMF as per standard of care in clinical practice.
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9
percentage of participants | 13.2 | 8.7 | 20.0 | 5.2 | 22.2

2. Secondary Outcome: Change From Baseline in the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: The CR-SMFRS is based on the investigator's clinical evaluation of the participant's chin and neck area using a 5-point ordinal scale (0 to 4) with 0=Absent Submental Convexity: no localized submental fat evident; 1=Mild Submental Convexity: minimal, localized submental fat; 2=Moderate Submental Convexity: prominent, localized submental fat; 3=Severe Submental Convexity; a marked amount of chin fat; and 4=Extreme Submental Convexity: marked, localized submental fat. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to the Follow-up Visit (Up to 9 Months) and Baseline to End of Treatment (EOT) Visit (Up to 18 Months)
Population: Full Analysis Set included all enrolled participants with a baseline visit and at least one post-baseline visit. Participants may have received more than one treatment. Number analyzed is the number of participants with data available for this outcome measure at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Not Elected Treatment: All enrolled participants who did not elect to have treatment for SMF.
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
score on a scale
  Baseline: number analyzed (Participants) | 568 | 23 | 5 | 77 | 9 | 674
  Baseline | 2.0 (0.8) | 2.7 (0.8) | 3.2 (0.8) | 1.7 (0.8) | 1.8 (1.1) | 2.0 (0.8)
  Change to Follow-up Visit: number analyzed (Participants) | 406 | 21 | 5 | 49 | 5 | 483
  Change to Follow-up Visit | -0.4 (0.7) | -1.6 (1.1) | -2.0 (1.0) | -0.7 (0.7) | -0.4 (0.6) | -0.5 (0.8)
  Change to EOT Visit: number analyzed (Participants) | 379 | 17 | 2 | 49 | 5 | 449
  Change to EOT Visit | -0.8 (0.8) | -2.1 (1.0) | -2.5 (0.7) | -0.9 (1.0) | -0.2 (0.5) | -0.8 (0.9)

3. Secondary Outcome: Change From Baseline in Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0 to 4) with 0=No chin fat at all, 1=A slight amount of chin fat, 2=A moderate amount of chin fat, 3=A large amount of chin fat, and 4=A very large amount of chin fat. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to the Follow-up Visit (Up to 9 Months) and Baseline to End of Treatment Visit (Up to 18 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
score on a scale
  Baseline: number analyzed (Participants) | 568 | 23 | 5 | 77 | 9 | 674
  Baseline | 2.0 (0.7) | 2.5 (0.7) | 3.2 (0.8) | 1.8 (0.7) | 2.0 (0.9) | 2.0 (0.7)
  Change to Follow-up Visit: number analyzed (Participants) | 409 | 21 | 5 | 48 | 5 | 485
  Change to Follow-up Visit | -0.3 (0.7) | -1.5 (0.9) | -2.2 (1.1) | -0.5 (0.8) | -0.8 (0.8) | -0.4 (0.8)
  Change to EOT Visit: number analyzed (Participants) | 383 | 17 | 2 | 49 | 4 | 452
  Change to EOT Visit | -0.7 (0.8) | -1.6 (0.9) | -2.0 (0.0) | -0.8 (0.9) | -0.5 (0.6) | -0.7 (0.8)

4. Secondary Outcome: Change From Baseline in the Patient-Reported Submental Fat Impact Scale (PR-SMFIS)
Description: The PR-SMFIS assesses the impact of submental fat on self-perception of 6 emotional and visual characteristics related to the appearance of submental fullness (unhappy, bothered, self-conscious, embarrassed, look older, and look overweight) as evaluated by the participant. Each item is rated on an 11-point numeric scale from 0 to 10. Scores for the 6 items were averaged to generate a PR-SMFIS total scale score ranging from 0 to 10 where 0 is a positive outcome and 10 is a negative outcome. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to the Follow-up Visit (Up to 9 Months) and Baseline to End of Treatment Visit (Up to 18 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
score on a scale
  Baseline: number analyzed (Participants) | 569 | 23 | 5 | 77 | 9 | 675
  Baseline | 6.9 (1.8) | 7.9 (1.5) | 9.0 (0.0) | 6.2 (2.2) | 7.0 (2.4) | 6.9 (1.9)
  Change to Follow-up Visit: number analyzed (Participants) | 408 | 21 | 5 | 48 | 5 | 484
  Change to Follow-up Visit | -1.2 (1.9) | -4.6 (2.3) | -6.6 (2.7) | -1.8 (2.4) | -2.4 (2.1) | -1.5 (2.2)
  Change to EOT Visit: number analyzed (Participants) | 382 | 17 | 2 | 49 | 4 | 451
  Change to EOT Visit | -2.8 (2.6) | -5.4 (2.6) | -6.5 (2.1) | -2.4 (2.7) | -2.3 (1.3) | -2.9 (2.7)

5. Secondary Outcome: Change From Baseline in the Subject Self Rating Scale (SSRS)
Description: The participant was asked to answer the question: "Considering your appearance in association with your face and chin, how satisfied do you feel with your appearance at the present time?" using a 7-point scale: 0=Extremely dissatisfied, 1=Dissatisfied, 2=Slightly dissatisfied, 3=neither satisfied nor dissatisfied, 4=Slightly satisfied, 5=Satisfied, and 6=Extremely satisfied. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to the Follow-up Visit (Up to 9 Months) and Baseline to End of Treatment Visit (Up to 18 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
score on a scale
  Baseline: number analyzed (Participants) | 569 | 23 | 5 | 77 | 9 | 675
  Baseline | 2.3 (1.4) | 2.0 (1.6) | 1.4 (1.5) | 2.1 (1.4) | 2.6 (1.2) | 2.2 (1.4)
  Change to Follow-up Visit: number analyzed (Participants) | 407 | 21 | 5 | 48 | 5 | 483
  Change to Follow-up Visit | 1.0 (1.7) | 2.4 (1.9) | 3.6 (2.1) | 1.6 (1.8) | 1.2 (2.2) | 1.1 (1.8)
  Change to EOT: number analyzed (Participants) | 382 | 17 | 2 | 49 | 4 | 451
  Change to EOT | 2.0 (2.0) | 2.8 (2.3) | 4.5 (2.1) | 2.1 (1.9) | 1.3 (1.5) | 2.1 (2.0)

6. Secondary Outcome: Change From Baseline in the Patient Self-Perception of Age (SPA)
Description: The participant rated their facial age in years at Baseline and at the End of Treatment Visit by answering the question: How many years difference compare to your actual age? A negative number indicates younger and a positive number indicates older. A negative change from Baseline indicates an improvement.
Time Frame: Baseline (Day 1) to End of Treatment Visit (Up to 18 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
years
  Baseline: number analyzed (Participants) | 569 | 23 | 5 | 77 | 9 | 675
  Baseline | -1.4 (5.0) | 0.5 (4.3) | 3.0 (6.7) | -0.5 (4.1) | -0.6 (3.2) | -1.2 (4.9)
  Change to EOT Visit: number analyzed (Participants) | 382 | 17 | 2 | 49 | 4 | 451
  Change to EOT Visit | -1.5 (5.3) | -5.6 (6.2) | -10.0 (0.0) | -0.6 (3.1) | -0.8 (4.4) | -1.6 (5.3)

7. Secondary Outcome: Change From Baseline in the Submental Skin Laxity Scale (SMSLG)
Description: SMSLG assessment was based on clinical evaluation and palpation of the submental area. The SMSLG scale incorporates 3 features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds).
  Grade 1 (none): no or minimal superficial wrinkling, skin well apposed to deeper neck structures, no skin redundancy [no skin draping or skin sagging]; Grade 2 (mild): mild superficial wrinkling, skin well apposed to deeper neck structures, minimal skin redundancy [slight skin draping and sagging]; Grade 3 (moderate): may have mild to moderate superficial wrinkling, skin has mild to moderate separation from deeper neck structures, moderate skin redundancy [moderate skin draping and skin sagging]; Grade 4 (severe): mild to marked superficial wrinkling, loose skin separated from deeper neck structures, marked skin redundancy [marked skin draping and sagging]. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to the Follow-up Visit (Up to 9 Months) and Baseline to End of Treatment Visit (Up to 18 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | Not Elected Treatment
Number analyzed (Participants) | 570 | 23 | 5 | 77 | 9 | 676
score on a scale
  Baseline: number analyzed (Participants) | 569 | 23 | 5 | 77 | 9 | 675
  Baseline | 2.0 (0.8) | 2.2 (0.7) | 2.0 (0.7) | 2.1 (0.8) | 2.0 (0.7) | 2.0 (0.8)
  Change to Follow-up Visit: number analyzed (Participants) | 405 | 21 | 5 | 49 | 5 | 482
  Change to Follow-up Visit | -0.1 (0.7) | -0.6 (1.0) | -0.4 (1.1) | -0.4 (0.6) | -0.4 (0.6) | -0.2 (0.7)
  Change to EOT Visit: number analyzed (Participants) | 378 | 17 | 2 | 49 | 5 | 448
  Change to EOT Visit | -0.2 (0.7) | -0.6 (1.0) | -0.5 (0.7) | -0.3 (0.6) | -0.2 (0.5) | -0.3 (0.7)

ADVERSE EVENTS:
Time Frame: Up to 19 Months
Description: Safety Population included all participants who received at least one treatment. Participants may have received more than one treatment.
Groups:
- All Treated Participants: All participants who received treatment for SMF as per standard of care in clinical practice: ATX1-101, Surgical Procedures, Laser Liposuction, Energy Devices or Other Treatments.
Arm/Group | Deoxycholic Acid (ATX-101) | Surgical | Laser Liposuction | Energy Devices | Other Treatments | All Treated Participants
Serious Adverse Events (participants affected / at risk) | 0/570 | 0/23 | 0/5 | 0/77 | 0/9 | 0/676
Other Adverse Events (participants affected / at risk) | 75/570 | 2/23 | 1/5 | 4/77 | 2/9 | 81/676
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid (ATX-101) (N=570) | Surgical (N=23) | Laser Liposuction (N=5) | Energy Devices (N=77) | Other Treatments (N=9) | All Treated Participants (N=676)
Injection site swelling (General disorders) | 59 | 1 | 1 | 4 | 1 | 63
Injection site hypoaesthesia (General disorders) | 38 | 0 | 0 | 1 | 1 | 39
Injection site bruising (General disorders) | 37 | 1 | 0 | 0 | 0 | 38
Injection site pain (General disorders) | 18 | 0 | 1 | 0 | 0 | 19
Injection site nodule (General disorders) | 5 | 0 | 1 | 0 | 0 | 6
Application site ulcer (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 2 | 3
Injection site oedema (General disorders) | 8 | 0 | 0 | 0 | 0 | 8
Injection site discomfort (General disorders) | 4 | 0 | 0 | 0 | 0 | 4
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Injection site nerve damage (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Injection site scab (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Uncoded (General disorders) | 2 | 0 | 0 | 0 | 0 | 2 — Uncoded
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Investigator shall allow Sponsor not less than 45 days to review any manuscript and not less than 30 days to review any poster presentation, abstract or any other written or oral material which describes or discloses the Study results. Institution and Investigator agree that because the Study is part of a multi-center Study, any publication by Institution or Investigator of the Study Results shall not be made before the first multi-center publication of participating sites.